CLINICAL TRIAL: NCT04861207
Title: Assessment of Tolerance and Effectiveness of Total Body Irradiation and Cladribine Before Allogeneic Hematopoietic Cell Transplantation in Patients With Acute Myeloid Leukemia and Myelodysplastic Syndromes
Brief Title: Total Body Irradiation and Cladribine Before Allogeneic Hematopoietic Cell Transplantation in Patients With AML (Acute Myeloid Leukemia) and Myelodysplastic Syndromes
Acronym: CLARA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-NIO-0001
Record Dates: First submitted 2021-04-25; First posted 2021-04-27 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia Myelodysplastic Syndromes
MeSH Terms: interventions — Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cladribine (Experimental)
  Interventions: Drug: Cladribine

INTERVENTIONS:
Drug: Cladribine — The conditioning regimen used will be cladribine-based at a dose of 5 mg / m2 for 5 days (iv.) and total body irradiation at a total dose of 12 Gy in three fractions.

SUMMARY:
A single center, prospective, one arm clinical study to assess the tolerance and effectiveness of total body irradiation and cladribine in adult patients diagnosed with AML( acute myeloid leukemia) and myelodysplastic syndromes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years.
2. Patient is a candidate for allogeneic hematopoietic cell transplantation due to acute myeloid leukemia(intermediate or high risk acute myeloid leukemia in complete remission, low risk with positive Minimal residual disease) or high risk myelodysplastic syndrome.
3. Demonstration of chemosensitivity in the case of treatment regimens with cladribine in induction therapy.
4. Patient signed informed consent form prior to any study related screening procedures are performed.
5. Patient has Eastern Cooperative Oncology Group performance status score of 0 or 1.
6. Patient is a candidate for allogeneic hematopoietic cell transplantation from sibling or unrelated donor (full matched or 9/10 mismatched) or from haploidentical donor.

Exclusion Criteria:

1. Has received more than 1 allogeneic hematopoietic cell transplantation.
2. Presence of active uncontrolled infection (i.e. sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection).
3. Known active human immunodeficiency virus, hepatitis B virus or hepatitis C virus infection (positive polymerase chain reaction test) or risk of hepatitis B virus reactivation (Hepatitis B surface antigen positive).
4. Presence of active disease in acute myeloid leukemia patients.
5. History or current diagnosis for uncontrolled or significant cardiac or pulmonary disease.
6. Presence of severe renal or liver dysfunction (creatinine, alanine aminotransferase,aspartate aminotransferase or bilirubin concentration > 3.0 upper limit of normal
7. Currently pregnancy or breast feeding.
8. Treatment of any other investigational agent in the same time as this study.
9. Known allergies, hypersensitivity, or intolerance to cladribine or similar compounds.
10. Women of childbearing potential who do not agree to use two effective methods of contraception.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The probability of progression-free survival in 24 month follow up | 24 month follow up

SECONDARY OUTCOMES:
Frequency of adverse events | 24 month follow up
24-month overall survival probability | 24 month follow up
Disease recurrence probability. | 24 month follow up
Mortality unrelated with disease recurrence | 24 month follow up
Likelihood of acute and chronic graft-versus-host disease | 24 month follow up
Time of neutrophil and platelet implantation | 24 month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Klinika Transplantacji Szpiku i Onkohematologii Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie Państwowy Instytut Badawczy, Oddział w Gliwicach, Gliwice, Poland